CLINICAL TRIAL: NCT01877330
Title: Intraplexus vs Extraplexus Injection of Local Anesthetic for Interscalene Block for Patients Undergoing Arthroscopic Shoulder Surgery
Brief Title: Optimal Location of Local Anesthetic Injection for Ultrasound Guided Interscalene Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISNB001
Record Dates: First submitted 2012-12-12; First posted 2013-06-13 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Shoulder Arthroscopy; Ultrasound-guided Interscalene Nerve Block
Keywords: shoulder arthroscopy; ultrasound guided nerve block; interscalene nerve block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injection in interscalene groove (Active Comparator): Patients undergoing shoulder arthroscopy will have an interscalene nerve block by injection of ropivacaine in the interscalene groove anterior and posterior to the brachial plexus nerves.
  Interventions: Procedure: Interscalene block for shoulder arthroscopy
- Injection between nerve roots (Active Comparator): Patients undergoing shoulder arthroscopy will have an interscalene nerve block by injection of ropivacaine in the interscalene groove inbetween the C5 and C6 nerve roots.
  Interventions: Procedure: Interscalene block for shoulder arthroscopy

INTERVENTIONS:
Procedure: Interscalene block for shoulder arthroscopy

SUMMARY:
This is a prospective randomized clinical trial to determine where is the optimal location for local anesthetic injection for ultrasound guided interscalene nerve blocks. The investigators are investigating if local anesthetic deposited between the nerve roots is more effective than local anesthetic deposited in the interscalene groove.

ELIGIBILITY:
Inclusion Criteria:

ASA I-II patients who are 18 years and older and who are scheduled for shoulder arthroscopy are eligible for enrollment provided they do not have any of the following exclusion criteria.

Exclusion Criteria:

* chronic pain
* high preoperative opioid requirement
* age < 18 years old
* non-English speaking
* contraindication to regional anesthesia (allergy to local anesthetics, coagulopathy, severe thrombocytopenia, pre-existing neuropathy in operative limb, infection at puncture site)
* need for postoperative nerve function monitoring
* patient refusal
* dementia
* pulmonary disease or low baseline oxygen saturation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Onset of motor blockade | 1 hour from time of injection
  Time to loss of shoulder abduction.

SECONDARY OUTCOMES:
Patient Satisfaction Score | 24 hours
Opioid consumption | 24 hours
  Opioid consumption - perioperative and post discharge
Quality of Nerve block | 24 hours
  onset of sensory block
Incidence of post-operative nausea/vomiting | 24 hours
Duration of nerve block | 24 hours
  Duration of analgesia from nerve block
Number of needle passes | 1 hour
Number of paresthesias | 1 hour
  number of paresthesia experience during nerve block
Residual paresthesia | 24 hour
  incidence of residual paresthesias

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Aleshi, MD, Principal Investigator — University of California, San Francisco; Monica W Harbell, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Orthopedic Institute, San Francisco, California, United States